CLINICAL TRIAL: NCT04974372
Title: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Brief Title: A Multicenter Clinical Study of Ultrasound Multimodal Imaging in the Evaluation of Heart Transplantation
Acronym: HT
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Xie Mingxing (Other)
Collaborators: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other); Shanghai Zhongshan Hospital (Other); Henan Provincial People's Hospital (Other); Wuhan Asia Heart Hospital (Other); Guangdong Provincial People's Hospital (Other)
Responsible Party: Sponsor-Investigator, Xie Mingxing, Department of Ultrasound, Union Hospital, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Organization: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Other Study IDs: 2021V1.0
Record Dates: First submitted 2021-07-10; First posted 2021-07-23 (Actual); Last update posted 2021-07-23 (Actual); Status verified 2021-07

CONDITIONS: Heart Transplant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- HT group: Patients have echocardiography examination before and after heart transplantation.
- Control group: healthy volunteers who had no history of hypertension, diabetes mellitus, renal failure or other organic diseases based on physical examinations, biochemical tests, electrocardiogram, echocardiography were enrolled as control group

SUMMARY:
The aims of this study are to 1. Assess the preoperative and postoperative atrial and ventricular structure and function comprehensively in heart transplantation; 2. Explore the early, accurately and non-invasively indicators for evaluating myocardial fibrosis in end-stage heart failure, as well detecting acute rejection (AR),coronary allograft vasculopathy(CAV) and adverse clinical events in heart transplant patients by using conventional and the advanced echocardiography.

DETAILED DESCRIPTION:
This study will enrolled 1000 HT patients and 500 healthy controls, and the cardiac structure and function will be evaluated by ultrasound multimodal imaging. And the study aimed to 1. Assess the preoperative and postoperative atrial and ventricular structure and function comprehensively in heart transplantation; 2. Explore the early, accurately and non-invasively indicators for evaluating myocardial fibrosis in end-stage heart failure, as well detecting acute rejection(AR),coronary allograft vasculopathy(CAV) and adverse clinical events in heart transplant patients by using conventional and the advanced echocardiography.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteers

Exclusion Criteria:

* had history of hypertension, diabetes mellitus, renal failure or other organic diseases based on physical examinations, biochemical tests, electrocardiogram, echocardiography

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: ALL adult HT recipients were consecutive prospectively enrolled who underwent transthoracic echocardiography (TTE) for surveillance at their routine follow-up visits at our institution
Sampling Method: Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2021-08-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Using Image-Pro Plus 6.0 software to measure myocardial fibrosis | the measurement of myocardial fibrosis up to 1 year after heart transplant
  The extent of myocardial fibrosis of the myocardial tissue from the removed heart during heart transplant was measured by Image-Pro Plus 6.0 software up to 1 year after heart transplant
All cause death after the inclusion of the study | All cause death happened after inclusion of this study, up to 5 years
  All cause death after HT was obtained via telephone interview with family members; contact with his/her physicians; or hospital records every year
Acute rejection after the inclusion of the study | Acute rejection happened after inclusion of this study, up to 5 years
  Acute rejection after the inclusion of the study was obtained at regular intervals via telephone interview with the patient, or if deceased, with family members; contact with his/her physicians; or hospital records every year
Cardiac allograft vasculopathy after the inclusion of the study | Cardiac allograft vasculopathy happened after inclusion of this study, up to 5 years
  Cardiac allograft vasculopathy after the inclusion of the study was obtained at regular intervals via telephone interview with the patient, or if deceased, with family members; contact with his/her physicians; or hospital records every year

SECONDARY OUTCOMES:
Major adverse cardiac events after the inclusion of the study | Major adverse cardiac events happened after inclusion of this study，up to 5 years
  Major adverse cardiac events after the inclusion of the study was obtained at regular intervals via telephone interview with the patient, or if deceased, with family members; contact with his/her physicians; or hospital records every year

CONTACTS AND LOCATIONS:
Overall Officials: Li Zhang, PhD, Principal Investigator — Department of Ultrasound, Union Hospital, Wuhan, China

IPD SHARING:
Plan to Share IPD: No